CLINICAL TRIAL: NCT04354974
Title: Evaluation of a Cognitive Remediation Program for Mood Disorders
Acronym: ECO-DBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Clémence ISAAC, clinical research unit director, Centre hospitalier de Ville-Evrard, France
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 10477M-ECO-DBP-2019
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Taking Charge of Cognitive Impairment in Patients With Mood Disorders

STUDY DESIGN:
Intervention Model Description: Evaluation of the specific therapeutic efficacy of Cognitive Training Therapy for Bipolar Patients on cognitive deficits in patients with bipolar disorder, treated over three months and followed up over nine months. Randomized, double-blind study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eco Program (Ecological Cognitive Training for Mood Disorders) (Active Comparator): Duration: four months, 16 sessions
  * Frequency: One one-hour session and one hour of personal work per week
  * Modalities: Paper and pencil exercises and manipulable tools
  * Objective: Learning problem-solving strategies for use in daily life
  * Modules: Psychoeducation, Information Processing, Memory, Concept Formation, Functional Disorders
  Interventions: Behavioral: Evaluation
- ThOR Program (Remission Oriented Therapy) (Active Comparator): Duration: four months, 16 sessions
  * Frequency: One one-hour session and one hour of personal work per week
  * Modalities: Paper tools and verbal exchange with the patient
  * Objective: Improvement of the patient's quality of life
  * Themes: Mood, social skills, autonomy, motivation, sleep
  Interventions: Behavioral: Evaluation

INTERVENTIONS:
Behavioral: Evaluation — Evaluation of a cognitive remediation program for mood disorders

SUMMARY:
Psychotherapeutic management of cognitive disorders in patients suffering from a mood disorder

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years old
2. The patient's previous diagnosis of Bipolar-Related Disorder or Depressive Disorder according to the DSM-5 criteria.
3. Mood stabilized with respect to depressive symptomatology (absence or presence of residual mild depressive symptoms (HDRS-17 ≤ 18))
4. Mood stabilized with respect to manic symptomatology (absence or presence of residual mild manic symptoms (YMRS ≤ 8))
5. Stable and effective treatment at minimum dose for at least 2 months
6. Cognitive complaint expressed by the patient, and detected by the patient's referring psychiatrist
7. Free and Informed Consent Form read, initialled and signed
8. Patient affiliated to a social protection scheme or beneficiary of State Medical Aid
9. Patient knowing how to speak French -

Exclusion Criteria:

1. Presence of a DSM-5 disorder, other than a mood, anxiety or personality disorder
2. Substance addiction or abuse (Alcohol, psychoactive substances) in the past 12 months
3. Manic, hypomanic or major depressive episode in the last 2 months
4. Somatic or neurological disorder which may lead to cognitive impairment
5. Current or less than one month's commitment to another research protocol
6. A neuropsychological assessment prior to 6 months.
7. Patient under protective custody, guardianship or reinforced guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-10-18 (Actual); Primary Completion 2022-02-18 (Estimated); Study Completion 2023-02-18 (Estimated)

PRIMARY OUTCOMES:
the Perceptual Reasoning Index (PRI) the Wechsler Intelligence Scale. | at 1 year
  Increase in the Perceptual Reasoning Index (PRI) of the Wechsler Adult Intelligence Scale - Fourth Edition [WAIS-IV] significantly different between the two study groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Youcef Bencherif, Neuilly-sur-Marne, France

IPD SHARING:
Plan to Share IPD: Yes